CLINICAL TRIAL: NCT01977768
Title: Phase III and Dose Ranging Trial of Heat-killed M. Vaccae (V7)
Brief Title: TB Immunotherapy Trial With Heat-killed M. Vaccae
Acronym: imm03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Immunitor LLC (Industry)
Collaborators: National Medical University, Ukraine (Other); Immunitor USA Inc. (Industry); University of Stellenbosch (Other); Lisichansk Regional Tuberculosis Dispensary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: imm03; imm03 (Other: immunitor)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Tuberculosis
Keywords: M. vaccae; TB; MDR-TB; V7-immunitor
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V7: Heat-inactivated M. vaccae pill (Experimental): Daily pill of V7 together with standard tuberculosis therapy
  Interventions: Biological: V7
- Placebo pill (Placebo Comparator): one pill of placebo pill once per day together with standard of care TB drugs
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V7 — One pill of V7 once daily for 30 days together with standard of care TB drugs
  Other Names: V7 or tableted heat-inactivated mycobacterium vaccae
  Arms: V7: Heat-inactivated M. vaccae pill
Biological: Placebo
  Arms: Placebo pill

SUMMARY:
The purpose of the study is to carry out multi-country (Ukraine and Mongolia), placebo-controlled, randomized Phase III trial in patients with drug-sensitive, multi-drug resistant (MDR-TB) and TB-HIV and identify efficacy and safety of whole-cell, heat-killed Mycobacterium vaccae formulated as a pill (V7) and consequently conduct confirmatory trials in intended registration countries, such as China, Russia and South Africa, etc.

DETAILED DESCRIPTION:
Main end-point is negative sputum conversion rate after one month in patients on V7 vs placebo arm, both arms will receive conventional anti-tuberculosis chemotherapy consisting of 1st and/or 2nd line TB drugs according to baseline diagnosis

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of TB
* sputum smear positive

Exclusion Criteria:

* pregnant
* likely to be non-compliant due to drug and/or alcohol abuse
* mentally unfit to comply with treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
bacillary sputum smear clearance | two years
  blinded assessment of sputum clearance score

SECONDARY OUTCOMES:
changes in body weight | 2 years
  comparison of body weight between treatment arm and placebo
changes in body mass index (BMI) | 2 years
  comparison of body mass index (BMI) between treatment arm and placebo
changes in inflammation markers | 2 years
  changes in erythrocyte sedimentation (ERS) rate and leukocyte counts
changes in liver function test | 2 years
  changes in ALT, AST and total bilirubin levels

OTHER OUTCOMES:
Immune correlates | 2 years
  Identify changes in immune cells (lymphocytes) resulting from V7 administration

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, PhD, MD/PhD, Principal Investigator — Immunitor LLC
Locations (2):
- Misheel Lung surgery hospital,, Ulaanbaatar, Ulaanbaatar, Mongolia
- Lisichansk Regional TB Dispensary, Lisichansk, Ukraine

REFERENCES:
- [Background] Butov DA, Efremenko YV, Prihoda ND, Zaitzeva SI, Yurchenko LV, Sokolenko NI, Butova TS, Stepanenko AL, Kutsyna GA, Jirathitikal V, Bourinbaiar AS. Randomized, placebo-controlled Phase II trial of heat-killed Mycobacterium vaccae (Immodulon batch) formulated as an oral pill (V7). Immunotherapy. 2013 Oct;5(10):1047-54. doi: 10.2217/imt.13.110. PMID 24088075
- [Background] Efremenko YV, Butov DA, Prihoda ND, Zaitzeva SI, Yurchenko LV, Sokolenko NI, Butova TS, Stepanenko AL, Kutsyna GA, Jirathitikal V, Bourinbaiar AS. Randomized, placebo-controlled phase II trial of heat-killed Mycobacterium vaccae (Longcom batch) formulated as an oral pill (V7). Hum Vaccin Immunother. 2013 Sep;9(9):1852-6. doi: 10.4161/hv.25280. Epub 2013 Jun 19. PMID 23782489
- [Background] Bourinbaiar AS, Mezentseva MV, Butov DA, Nyasulu PS, Efremenko YV, Jirathitikal V, Mishchenko VV, Kutsyna GA. Immune approaches in tuberculosis therapy: a brief overview. Expert Rev Anti Infect Ther. 2012 Mar;10(3):381-9. doi: 10.1586/eri.12.1. PMID 22397570
- [Result] Atmakuri K, Penn-Nicholson A, Tanner R, Dockrell HM. Meeting report: 5th Global Forum on TB Vaccines, 20-23 February 2018, New Delhi India. Tuberculosis (Edinb). 2018 Dec;113:55-64. doi: 10.1016/j.tube.2018.08.013. Epub 2018 Aug 24. PMID 30514514
- [Derived] Bourinbaiar AS, Batbold U, Efremenko Y, Sanjagdorj M, Butov D, Damdinpurev N, Grinishina E, Mijiddorj O, Kovolev M, Baasanjav K, Butova T, Prihoda N, Batbold O, Yurchenko L, Tseveendorj A, Arzhanova O, Chunt E, Stepanenko H, Sokolenko N, Makeeva N, Tarakanovskaya M, Borisova V, Reid A, Kalashnikov V, Nyasulu P, Prabowo SA, Jirathitikal V, Bain AI, Stanford C, Stanford J. Phase III, placebo-controlled, randomized, double-blind trial of tableted, therapeutic TB vaccine (V7) containing heat-killed M. vaccae administered daily for one month. J Clin Tuberc Other Mycobact Dis. 2019 Dec 12;18:100141. doi: 10.1016/j.jctube.2019.100141. eCollection 2020 Feb. PMID 31890902